CLINICAL TRIAL: NCT00805857
Title: SCOLTA: SURVEILLANCE COHORT LONG-TERM TOXICITY ANTIRETROVIRALS
Brief Title: Surveillance Cohort Long-term Toxicity Antiretrovirals in HIV-infected Patients Enrolled in TPV Cohort
Status: Withdrawn | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1182.144
Record Dates: First submitted 2008-06-10; First posted 2008-12-10 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

INTERVENTIONS:
Drug: Tipranavir

SUMMARY:
The SCOLTA project is a system for online surveying of adverse events to recently commercialized antiretroviral drugs and a sentinel for unexpected and late adverse events reactions arising during any antiretroviral treatment.Aim of the proposed study is:

1. to evaluate the prevalence and incidence of serious adverse events and serious unexpected adverse events in HIV-infected patients enrolled in the SCOLTA project Tipranavir cohort and to identify possible risk factors
2. the evaluation of tipranavir containing regimens durability, considering treatment interruption for each reason.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 years old HIV infected treated with tipranavir

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prevalence and incidence of serious adverse events and serious unexpected adverse events in HIV infected patients enrolled in Tipranavir cohort and to identify possible risk factors | 48wks

SECONDARY OUTCOMES:
the evaluation of tipranavir containing regimens durability, considering treatment interruption for each reason | 48wks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim